CLINICAL TRIAL: NCT03243955
Title: Transcutaneous Electrical Acupoint Stimulation (TEAS) for Chronic Constipation
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Andrew Shubov, MD, Principal Investigator, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 441356-KH-50890
Record Dates: First submitted 2017-05-02; First posted 2017-08-09 (Actual); Last update posted 2023-10-03 (Actual); Status verified 2023-10

CONDITIONS: Constipation - Functional
Keywords: acupuncture; TENS; TEAS; constipation; transcutaneous
MeSH Terms: conditions — Constipation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: the patient is unaware which group he is assigned to the researchers discussing this with the patients are unaware of group assignment the investigator is unaware of group assignment the outcomes assessor is unaware of group assignment until data analysis is complete
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- TEAS (Active Comparator): True acupoint locations for placement of TENS unit pads
  Interventions: Device: Verum TEAS
- Placebo (Sham Comparator): non-acupoint locations for placement of TENS unit pads
  Interventions: Device: Sham TEAS

INTERVENTIONS:
Device: Verum TEAS — TENS unit with electrodes applied to acupuncture point locations
  Arms: TEAS
Device: Sham TEAS — TENS unit with electrodes applied to non-acupuncture point locations
  Arms: Placebo

SUMMARY:
Transcutaneous electrical acupoint stimulation (TEAS) is an emerging technology for non-invasive neuromodulation that has broad potential implications and warrants further study. The investigators' clinical experience from the University of California, Los Angeles (UCLA) Center for East-West Medicine (CEWM) has also demonstrated that TEAS can be used as an effective self-care tool for patients with chronic illness who do not have the time or resources for frequent acupuncture treatments. Chronic constipation is the chosen area of study because of the large population with a substantial impairment in health-related quality of life and work productivity. The investigators have recently completed a randomized controlled trial (RCT) demonstrating the benefit of perineal self-acupressure on quality of life measurements in this population, which supports investigation into other acupuncture-based self-care interventions. Given these findings, the investigators hypothesize that home patient-administered TEAS can provide measurable improvements in both symptom severity and health related quality of life.

DETAILED DESCRIPTION:
This study will be a double blinded randomized controlled trial. Respondents will be screened by phone and qualified subjects will be sent home for 2 weeks to complete a bowel movement logbook, then return into the CEWM office where they will submit validated surveys (specifically, the PAC-SYM and PAC-QOL) and have a photo taken of their tongue. A baseline non-invasive heart rate variability (HRV) measurement will be taken at this time as well. Study personnel will instruct each subject on TEAS pad placement and how to use the device, but not tell the subjects where to place the pads. The subjects will been assigned to one of two experimental groups (verum and sham) based on a 1:1 random allocation, with the study personnel blinded to the allocation. Both groups will be given transcutaneous electrical nerve stimulator (TENS) units with pre-set parameters and access to the adjustable amplitude dial for self-adjustment of amplitude, with the verum group given pre-printed information on proper application on true acupoints, and sham group will be given information on non-acupuncture points. The subjects will be instructed on daily use for 30 minutes per day for at least 5 days per week, and asked to track device use as well as bowel movement frequency and quality using a logbook. They will also submit to an online survey every week during the 4-week trial period. At the conclusion of the study, they will return the units and repeat the survey and HRV measurements.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Satisfy a modified ROME-IV criteria for functional constipation including:

  * Fewer than three spontaneous bowel movements per week
  * and meet one of the following symptoms for at least 12 weeks in the preceding 12 months:

    * straining during >25% of the bowel movements (BMs)
    * lumpy or hard stools during >25% of BMs
    * sensation of incomplete evacuation during >25% of BMs
    * sensation of anorectal obstruction or blockage for >25% of BMs
    * manual maneuvers to facilitate >25% of BMs
  * loose stools are rarely present without the use of laxatives
  * insufficient criteria for IBS (does not have recurrent abdominal pain at least 1 day per week in the past 3 months)
* able to understand and provide written consent
* If over age 50, have undergone routine colon cancer screening (colonoscopy, sigmoidoscopy, colonography or fecal occult blood testing)
* subjects must have normal serum chemistry and normal thyroid stimulating hormone (TSH) within the past year
* subjects must have normal sensation over the areas where the pads will be placed (lumbar region and lower extremities surrounding the knees anteriorly)

Exclusion Criteria:

* Pregnancy
* Numbness around the genitals or groin, bladder or bowel dysfunction or incontinence, new sciatica type leg pain or new onset sexual dysfunction within the past year.
* Any changes to constipation related medications over the past 1 month
* Use of rescue medication (polyethylene glycol, bisacodyl, enema, etc) greater than once per week
* Pacemaker, implanted cardiac defibrillator or other implanted electrical device
* 10% weight loss in past 6 months
* New onset Hematochezia since last medical evaluation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2017-02-28 (Actual); Primary Completion 2025-07-01 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
spontaneous bowel movement (SBMs) per week | 4 weeks
  Comparison of weekly spontaneous bowel movement (SBMs) per week between the two groups using a paired t-test comparing the final time point to the lead-in measurement.

SECONDARY OUTCOMES:
Responder rate | 4 weeks
  Comparison of the responder rate (responder defined as having >1 SBM per week for 2 out of the 4 treatment weeks) at the end of the study in each group
PAC-QOL | 4 weeks
  Paired t-test will be used to compare the average PAC-QOL scores between baseline and final measurements
PAC-SYM | 4 weeks
  Paired t-test will be used to compare the average PAC-SYM scores between baseline and final measurements
HRV Changes | 4 weeks
  Comparison of the differences between the high frequency (HF), low frequency (LF), and LF/HF measures of the spectral analysis of HRV (heart rate variability) between the baseline and study conclusion
Bristol Stool Scale | 4 weeks
  Comparison of the differences in the average Bristol Stool Scale between the baseline and study conclusion

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Shubov, MD, Principal Investigator — University of California, Los Angeles
Locations (1):
- University of California, Los Angeles, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No